CLINICAL TRIAL: NCT06315790
Title: Safety and Efficacy of Botulinum Toxin A in Patients With Trigeminal Neuralgia: a Double-blind, Randomized, Placebo-controlled, Parallel-group Trial and Investigation of Neuro-inflammatory Biomarkers as Predictors of Efficacy
Brief Title: Safety and Efficacy of Botulinum Toxin A in Patients With Trigeminal Neuralgia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henrik Schytz (Other)
Responsible Party: Sponsor-Investigator, Henrik Schytz, Consultant, Associate Professor, DMSc, PhD, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TN BTX-A Trial
Record Dates: First submitted 2023-08-28; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isotonic saline (Placebo Comparator)
  Interventions: Other: Isotonic saline
- Botulinum toxin A (Active Comparator)
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — Subcutaneously injections are given unilaterally in the face at predefined injection sites.
  Arms: Botulinum toxin A
Other: Isotonic saline — Subcutaneously injections are given unilaterally in the face at predefined injection sites.
  Arms: Isotonic saline

SUMMARY:
This is a double-blind randomized clinical trial comparing the pain reduction of individuals treated with BTX-A and placebo as well as evaluating possible changes in neuroinflammatory biomarkers. The trial lasts 16 weeks, with a 4-week baseline phase and a 12-week randomization phase. Four visits are planned: 1) Introduction and baseline data collection, 2) Medical evaluation and treatment assignment, 3) Follow-up with biomarker analysis, and 4) Trial conclusion interview. 80 participants will be included and randomized 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of classical TN or idiopathic TN according to criteria of The International Classification of Headache Disorders 3rd edition.
2. Age between 18 and 85 years.
3. Subjects must experience pain defined as a minimum of three TN related pain paroxysms per day at least four days a week of an average intensity of 4 to 10, inclusive, on the 11-point NRS (0 = no pain; 10 = maximum pain imaginable) during the last 4 weeks to enter the baseline phase.
4. During baseline phase subjects must experience pain defined as a minimum of three TN related pain paroxysms per day at least four days a week of an intensity of an average 4 to 10, inclusive, on the 11-point NRS (0= no pain; 10= maximum pain imaginable) during the last month to enter the treatment phase (to be randomized).
5. Fluency in Danish.

Exclusion Criteria:

1. Severe cardiovascular and cerebrovascular disease such as ischemic heart disease, myocardial infarction or previous stroke or transient ischemic attack, major CVD interventions during the last three months.
2. Expected poor compliance, i.e., considered unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge.
3. Ongoing and unstable severe psychiatric disease.
4. Anamnestic or clinical symptoms of any kind that are deemed relevant for study participation by the physician who examines the patient.
5. Change of TN treatment or treatment dose within two weeks prior to the baseline visit.
6. Previous treatment with BTX-A for facial pain.
7. Loading treatment within 4 weeks with phenytoin or sodium valproate.
8. Female subjects either pregnant, breastfeeding or with planned conception within the study period.
9. Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during the study.
10. Known allergy to any component of BTX-A.
11. Infection at the proposed injection site.
12. Known severe neuromuscular disorders or any degree of disorder affecting the neuromuscular transmission.
13. Known comprised respiratory function.
14. Member of investigational site staff or relative of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders in botulunim toxin A and placebo group | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Responders are participants with a 30 % reduction in mean average daily pain score.

SECONDARY OUTCOMES:
Biomarkers | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  The degree of concentration change in inflammatory biomarkers (CGRP, CRP, TNF alpha, IL1, IL2, and IL6) in responders versus non-responders in BTX-A and placebo group.
Tear fluid CGRP | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  The difference in tear fluid calcitonin gene-related peptide (CGRP) between the symptomatic side and the asymptomatic side.
50 % reduction | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  The proportion of subjects reaching ≥50% reduction in mean Average Daily Pain (ADP) intensity score
75 % reduction | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  The proportion of subjects reaching ≥75% reduction in mean ADP
Prolonged 30 % reduction | Week 9 to 12 compared with baseline (week -4 to -1)
  The proportion of subjects reaching ≥30% reduction in mean ADP
Change in paroxysms | Evaluation period (week 2 to 5) and during weeks 9 to 12 compared with baseline (week -4 to -1)
  Change in mean number of daily pain paroxysms n BTX-A group and placebo group
PGI-C | Week 5
  Proportion of subjects with a Patient Global Impression of Change (PGI-C) scale response of "much improved" or "very much improved" in BTX-A and placebo group
PENN Facial Pain Scale-Revised (PENN-FPS-R) | Baseline to week 5
  Change in the PENN-FPS-R
Patient's guess | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Proportion of subjects correctly guessing whether they received BTX-A or placebo
Dropouts | Up to 24 weeks
  Proportion of dropouts caused by increased intake of trigeminal neuralgia (TN) medication or use of rescue medication in BTX-A group compared to the placebo group through study completion.
Side effects | Up to 24 weeks
  Proportion of subjects with side-effects registered in weeks 2 to 5 during treatment with BTX-A compared with placebo through study completion.

OTHER OUTCOMES:
Pure paroxysmal pain vs. paroxysms with concomitant pain | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Patients with purely paroxysmal pain versus patients with concomitant continuous pain.
Idiopathic vs. classical trigeminal neuralgia | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Patients with idiopathic trigeminal neuralgia versus patients with classical trigeminal neuralgia
Patients with severe pain | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Patients with severe pain (defined as ADP ≥7 ) versus patients with less severe pain (ADP < 7)
Gender distribution | Evaluation period (week 2 to 5) compared with baseline (week -4 to -1)
  Male patients versus female patients
Disease duration | Baseline
  Patients with a long duration of TN (≥ 5 years) versus patients with a short duration of TN (< 5 years).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No